



Sub-study: The effect of prior exposure to the Measles, Mumps and Rubella vaccine on innate and adaptive immune responses to a SARS-CoV-2 mRNA vaccine

# STATISTICAL ANALYSIS PLAN

VERSION 1.2, 21 September 2021

Protocol version Clinicaltrials.gov

2.0 dated 28 Feb 2021 NCT04646239



# **Table of contents**

| ABBR | EVIATIONS | 3 |
|-------------------|------------------------------------|----------------|
| LIST C | OF AUTHORS AND REVIEWERS | 4 |
| 1 | INTRODUCTION | 5 |
| 1.1<br>1.2<br>1.3 | , | 5 |
| 2 | STUDY METHODS | |
| 2.1<br>2.2<br>2.3 | | 7 |
| 2.4 | | |
| 2.5 | Study outcomes | 8 |
| 3 | STATISTICAL PRINCIPLES | 9 |
| 3.1<br>3.2 | | 9 |
| 3.3 | | |
| | 3.3.1 Adjustment factors | |
| | 3.3.3 Secondary endpoints analysis | |
| 4 | REFERENCES ERROR! BOOKMAR | K NOT DEFINED. |
| 5 | APPROVALS | 11 |
| 6 | REVISION HISTORY | 12 |



# **ABBREVIATIONS**

| AE | Adverse Event |
|------------|-----------------------------------------------|
| BCG | Bacille Calmette-Guerin |
| CCTU | Comprehensive Clinical Trials Unit |
| COVID-19 | SARS-CoV-2-induced disease |
| DMC | Data Monitoring Committee |
| EC50 | Half-maximum effective concentration |
| IC50 | Half-maximum inhibitory concentration |
| IFN | Interferon |
| IL | Interleukin |
| ITT | Intention-To-Treat |
| MMR | Measles, Mumps and Rubella vaccine |
| NK | Natura Killer |
| OPV | Oral Polio Vaccine |
| OR | Odds Ratio |
| PCR | Polymerase Chain Reaction |
| RPMI | Roswell Park Memorial Institute |
| SAE | Serious Adverse Event |
| SARS-CoV-2 | Virus causing COVID-19 |
| SUSAR | Suspected Unexpected Serious Adverse Reaction |
| TNF | Tumor Necrosis Factor |
| TSC | Trial Steering Committee |
| UCL | University College London |
| WHO | World Health Organisation |



#### LIST OF AUTHORS AND REVIEWERS

#### **Author**

Dr Hakim-Moulay Dehbi, lead trial statistician, Comprehensive Clinical Trials Unit (CCTU), University College London (UCL), United Kingdom (UK)

#### **Reviewers**

Professor Michael Avidan, Clinical Coordinating Centre Principal Investigator, Washington University School of Medicine in St Louis, USA

Dr Leon du Toit, Anaesthesiologist at Washington University School of Medicine in St Louis, USA

Professor Mihai Netea, Infectious Diseases Specialist, Radboud University Medical Center in Nijmegen, The Netherlands.



#### 1 INTRODUCTION

## 1.1 General principles of the Statistical Analysis Plan (SAP)

This document details the proposed analysis strategy for the sub-study of CROWN CORONATION, leading to scientific publication(s). The results reported in these papers will follow the strategy set out here, which adheres to the guidelines for the content of a statistical analysis plan<sup>1</sup>. Moreover, the reporting of the main trial will adhere to the CONSORT guidelines<sup>2</sup>.

Suggestions for subsequent analyses by oversight committees, journal editors or referees, will be considered carefully in line with the principles of this analysis plan. Subsequent analyses of a more exploratory nature will not be bound by this strategy, and will be detailed in separate analysis plans.

Any deviations from the SAP will be described and justified in the final reports. This document is intended to be stand-alone from the protocol and adhere to the main points in the analysis summary specified in the protocol. However, the SAP can undergo revision outside of the protocol.

# 1.2 Background and rationale of the sub-study

Adaptive memory immune responses (particularly B cells and antibodies) are considered the cornerstone of vaccination in humans. However, recent studies demonstrate that a memory-like response in innate immunity can also enhance resistance to infection. These observations have led to the paradigm-shifting concept of trained immunity, where functional reprogramming of innate immune cells such as monocytes, macrophages, and Natural Killer (NK) cells can improve immune responses against infections. Epidemiological studies have shown that certain vaccines employing live attenuated microorganisms such as Bacille Calmette-Guerin (BCG), measles-containing vaccines (such as MMR), and oral polio vaccine (OPV) exert heterologous protective effects against infections other than those for which these vaccines are administered, and this cannot be explained by induction of any specific T- or B cell responses. Vaccination with measles seems to induce a transient suppression of lymphoproliferative responses, but an increase in innate immune responses, as measured by nonspecific cytokine production.

Recent exposure to a vaccine may affect the immune response to subsequent vaccination with an unrelated vaccine. Such interaction between different vaccines has not been studied extensively. Evidence suggests that the chronological order of different vaccines in childhood immunization schedules can have a notable impact on overall childhood mortality. Interaction between vaccines may occur through modification of the adaptive response and / or modification of the innate immune response. Such interaction can be either positive or negative.

The rapid development and roll-out of specific SARS-CoV-2 mRNA vaccination in the USA,



coincided with enrolment of participants into the CROWN CORONATION trial (NCT04333732) – a study investigating the efficacy of the MMR vaccine to prevent symptomatic, PCR positive COVID-19. Subsequent to randomization to either MMR or placebo injection, a number of participants in the CROWN CORONATION trial were vaccinated with a SARS-CoV-2 mRNA vaccine.

# 1.3 Objectives of the sub-study

The goal of this sub-study is to characterize and compare, in those exposed to a) recent MMR vaccination followed by SARS-CoV-2 vaccination and b) recent placebo injection followed by SARS-CoV-2 vaccination,

- I) the in-vitro, cytokine and chemokine responses (tumor necrosis factor (TNF)- $\alpha$ , interleukin (IL)-1 $\beta$ , IL-6, IL-10, IL-17, IL-22, interferon (IFN)- $\alpha$ , and IFN- $\gamma$ ) to heterologous stimuli.
- II) the SARS-CoV-2 neutralization assay (half-maximum effective concentration [EC50]; half-maximum inhibitory concentration [IC50]).



#### **2 STUDY METHODS**

#### 2.1 Trial design

This is a sub-study within the CROWN CORONATION trial.

At Washington University in St Louis, consenting participants are recruited into the sub-study. Additional blood samples will be required from participants in the sub-study, to enable measurement of the outcomes of the sub-study. Apart from additional blood samples that will be collected from those in the sub-study, these participants will be treated the same as those taking part in the CROWN CORONATION trial.

#### 2.2 Framework

CROWN CORONATION is a superiority trial. The aim is to demonstrate that the trial intervention(s) is(are) effective at decreasing the incidence of symptomatic COVID-19 disease.

In the sub-study, we hypothesize that, compared to SARS-CoV-2 mRNA vaccination alone, MMR vaccination prior to SARS-CoV-2 mRNA vaccination will induce lasting trained immunity in recipients, manifested by improved innate immune responses upon in vitro exposure of supernatants to heterologous pathogen products. We also hypothesize that MMR vaccination prior to SARS-CoV-2 mRNA vaccination does not alter the adaptive immune response to SARS-CoV-2 mRNA vaccination.

#### 2.3 Randomisation

Sequence generation, allocation and implementation takes place within the CROWN CORONATION trial.

#### 2.4 Sample size

All CROWN CORONATION participants who meet the inclusion criteria will be contacted for recruitment. We will enrol as many participants as possible into the sub-study. The eligible population size is 160.

For the purpose of sample size calculation, we used the t-test to compare the primary outcome between treatment arms, i.e. the difference in cytokine and IFN- $\gamma$  response between MMR and placebo groups. Table 1 reports power given the expected difference in IFN- $\gamma$  responses, with a two-sided type-1 error rate of 5%.

Table 1: Predicted power.



| Stimulus | Expected difference between means (pg/ml) | Expected<br>standard<br>deviation | Power with<br>60<br>participants | Power with<br>100<br>participant<br>s | Power with<br>140<br>participant<br>s |
|---|---|---|---|---|---|
| TLR-3 ligand | 400 | 900 | 39% | 59% | 74% |
| TLR-7/8<br>ligand | 450 | 900 | 48% | 70% | 84% |

# 2.5 Study outcomes

- i) Primary outcomes:
  - a. PBMC cytokine production (TNF- $\alpha$ , IL-1 $\beta$ , IL-6, and IFN- $\alpha$ ) 1 day after stimulation with heterologous products (inactivated SARS-CoV-2, live attenuated MMR viruses, toll-like receptor (TLR)-3 ligand, TLR-7/8 ligand, TLR-4 ligand, and RPMI medium).
  - b. IL-10, IL-17, IL-22, and IFN-γ production 5 days after stimulation of PBMCs with heterologous products.
- ii) Secondary outcomes:
  - c. SARS-CoV-2 neutralization assay (EC50; IC50).
  - d. Measles IgG antibody titres

Timing: Blood collected at a single sub-study visit around 6 to 9 weeks following the participant's second SARS-CoV-2 mRNA vaccine injection.



#### **3 STATISTICAL PRINCIPLES**

This sub-study is hypothesis generating. No adjustment will be made for multiple testing. All results comparing the treatment arms will be provided with 95% confidence interval (except if specified otherwise). Analysis will be for complete cases; no imputation will be performed for missing data. Missing data will be summarised and reported with results.

# 3.1 Analysis population

All randomised participant data will be included in the Intention-To-Treat (ITT) analysis according to the arm they were randomised to, irrespective of the actual study drug that they took. This ITT analysis will be the main strategy for the sub-study (primary and secondary outcomes).

A modified ITT analysis will be performed at the end of the CROWN CORNATION trial, based on serology results. Participants with evidence of COVID-19 infection at the start of the study will be removed from the analysis set. It is anticipated that this sub-study will be completed and reported on prior to analysis of the main trial so that the modified ITT analysis of the substudy data will be reported separately.

### 3.2 Baseline patient characteristics

Baseline characteristics will be summarised for all participants in the sub-study. Summary measures for the baseline characteristics will be presented as mean and standard deviation for continuous (approximate) normally distributed variables, medians and interquartile ranges for non-normally distributed continuous variables, and frequencies and percentages for categorical variables. We will plot histograms of continuous variables to assess normality.

#### 3.3 Analysis methods

The results of the analyses will be reported following the principle of the ICH E3 guidelines on the Structure and Content of Clinical Study Reports<sup>5</sup>. There will be no imputations for missing data.

Endpoints will be summarised graphically with box-whisker-dot plots.

#### 3.3.1 Adjustment factors

All models for the primary outcomes will be adjusted for sex and the calendar date of sample collection (by quarter of the year). Diagnostics for regression models will be assessed to ensure that underlying assumptions are met.

Sensitivity analyses will be performed by individually adding adjustment for age, interval duration between last SARS-CoV-2 vaccine injection and blood draw, interval duration between MMR or placebo injection and blood draw, and interval duration between MMR or



placebo injection and SARS-CoV-2 vaccination (figure 1). Outcomes will be plotted over time to assess the effect of the stated interval durations (figure 1) on the measured outcomes.



Figure 1: Interval durations in sub-study

#### 3.3.2 Primary endpoints analysis

TNF- $\alpha$ , IL-1 $\beta$ , IL-6, IL-10, IL-17, IL-22, IFN- $\alpha$  and IFN- $\gamma$  will be analysed by linear regression, with a coefficient for treatment arm, and adjusted for sex and the calendar date (which quarter of the year) of sample collection. The endpoints will be reported as the adjusted mean (95% CI) effect of MMR pre-exposure on the endpoint. For each specified endpoint, the individual participant assay response to RPMI will be evaluated and if the response is greater that three times the lower detectable limit of the assay, the data from that participant will be excluded from analysis for the specific endpoint. For example, if the IL-6 value is greater than three times the lower detectable limit in response to RPMI, the participant's data will be excluded from the analyses of IL-6 responses to the heterologous stimuli. The participant's data will still be used for the other endpoints in which the assay response to RPMI was less than three times the lower detectable limit.

#### 3.3.3 Secondary endpoints analysis

SARS-CoV-2 neutralization assay (EC50; IC50) and Measles IgG antibody titres will be analysed by linear regression, with a coefficient for treatment arm, and adjusted for sex and the calendar date (which quarter of the year) of sample collection.



# 4 APPROVALS

| Lead Trial<br>Statistician | Name: Hakim-Moulay Dehbi | |
|---|---|---|
| | Signature: | Date: 04 Oct 2021 |
| Investigator | Name: Leon du Toit | |
| | Signature: | Date: 30 Sep 2021 |



# **5 REVISION HISTORY**

| Version | Date | Edited<br>by | Comments/Justification | Timing in relation to first unblinded analysis |
|---|---|---|---|---|
| 0.1 | 27/07/2021 | HMD | First draft | Prior |
| 0.2 | 04/08/2021 | LDT | Revision | Prior |
| 1.0 | 10/08/2021 | LDT | Version 1 | Prior |
| 1.1 | 15/09/2021 | LDT | Revision | Prior |
| 1.2 | 21/09/2021 | HMD | Version 1.1 | Prior |